CLINICAL TRIAL: NCT00003425
Title: Phase I/II Study of Escalating Dose Melphalan With Autologous Pluripotent Hematopoietic Stem Cell Support and Amifostine Cytoprotection in Cancer Patients
Brief Title: Phase I/II Study of Escalating-Dose Melphalan w/Autologous SCS & Amifostine Cytoprotect
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Kentucky (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKMC-97BMT72; CDR0000066448 (Registry Identifier: PDQ (Physician Data Query)); ALZA-UKMC-97BMT72; NCI-V98-1455
Record Dates: First submitted 1999-11-01; First posted 2004-02-20 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Breast Cancer; Leukemia; Lymphoma; Neuroblastoma; Ovarian Cancer; Sarcoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer; recurrent adult Hodgkin lymphoma; refractory multiple myeloma; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; regional neuroblastoma; disseminated neuroblastoma; stage 4S neuroblastoma; recurrent neuroblastoma; stage III multiple myeloma; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; unspecified adult solid tumor, protocol specific; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; ovarian stromal cancer; stage III ovarian germ cell tumor; stage IV ovarian germ cell tumor; recurrent ovarian germ cell tumor; acute undifferentiated leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; secondary acute myeloid leukemia; borderline ovarian surface epithelial-stromal tumor; ovarian sarcoma; localized unresectable neuroblastoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Breast Neoplasms; Leukemia; Lymphoma; Neuroblastoma; Ovarian Neoplasms; Sarcoma; Hodgkin Disease; Multiple Myeloma; Carcinoma, Ovarian Epithelial; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Neuroectodermal Tumors, Primitive, Peripheral; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Filgrastim; Amifostine; Cyclophosphamide; Melphalan; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Amifostine trihydrate (Experimental)
  Interventions: Biological: filgrastim; Drug: amifostine trihydrate; Drug: cyclophosphamide; Drug: melphalan; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: amifostine trihydrate
  Other Names: WR-2721
Drug: cyclophosphamide
Drug: melphalan
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. Chemoprotective drugs such as amifostine may protect normal cells from the side effects of chemotherapy.

PURPOSE: Phase I/II trial to study the effectiveness of high-dose melphalan plus peripheral stem cell transplantation and amifostine in treating patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of high dose melphalan with autologous peripheral blood stem cell support and amifostine cytoprotection in patients with cancer. II. Determine the complete response rate, event free survival, overall survival, and nonrelapse mortality in this patient population.

OUTLINE: This is a dose escalation study of melphalan. Prior to high dose melphalan and amifostine cytoprotection, patients may receive cyclophosphamide IV. Filgrastim (G-CSF) is given until cytapheresis is completed. Patients receive high dose melphalan according to an escalating dose schedule. High dose melphalan is administered IV on day -1. Amifostine is also administered on days -2 and -1. Peripheral blood stem cell transplantation is performed on day 0. Dose escalation of high dose melphalan continues until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 8 patients experience dose limiting toxicity. After the MTD of high dose melphalan is determined, additional patients are treated at this dose level. Patients are followed at days 30, 100, 365, and yearly thereafter.

PROJECTED ACCRUAL: After the determination of MTD, a total of 14-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Confirmed diagnosis of primary tumor and/or recurrence that has a low curative potential using other therapies, including but not limited to: Acute leukemia Myeloma Breast cancer Ovarian cancer Hodgkin's disease Non-Hodgkin's lymphoma Neuroblastoma Ewing's sarcoma In the absence of recurrence, malignancies for which an autotransplant regimen is considered a reasonable therapeutic alternative are also considered Greater than 25% of bone marrow normal cellularity and less than 10% of volume composed of tumor cells No active brain metastases or carcinomatous meningitis (controlled CNS metastases eligible)

PATIENT CHARACTERISTICS: Age: 14 to 70 Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC greater than 3000/mm3 Absolute neutrophil count greater than 1500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin, SGOT, and SGPT less than 2 times normal Renal: Creatinine clearance greater than 60 mL/min Cardiovascular: LVEF at least 45% Pulmonary: DLCO at least 50% FEV1 at least 60% Other: Not pregnant or nursing Fertile patients must use effective contraception HIV, HTLV-1, and HTLV-2 negative Hepatitis B and C negative

PRIOR CONCURRENT THERAPY: Biologic therapy: No more than 1 prior autologous peripheral blood stem cell transplant Chemotherapy: Cumulative anthracycline or equivalent dose no greater than 450 mg/m2 Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: Recovered from prior therapy No antihypertensives during and 24 hours prior to amifostine administration

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 1997-12; Primary Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna E. Reece, MD, Study Chair — Lucille P. Markey Cancer Center at University of Kentucky
Locations (4):
- United States (4):
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Result] Phillips GL, Meisenberg BR, Reece DE, Adams VR, Badros AZ, Brunner JL, Fenton RG, Filicko J, Grosso DL, Hale GA, Howard DS, Johnson VP, Kniska A, Marshall KW, Mookerjee B, Nath R, Rapoport AP, Sarkodee-Adoo C, Takebe N, Vesole DH, Wagner JL, Flomenberg N. Activity of single-agent melphalan 220-300 mg/m2 with amifostine cytoprotection and autologous hematopoietic stem cell support in non-Hodgkin and Hodgkin lymphoma. Bone Marrow Transplant. 2004 Apr;33(8):781-7. doi: 10.1038/sj.bmt.1704424. PMID 14767498
- [Derived] Skliarova T, Lara-Cabrera ML, Hafstad H, Havnen A, Saether SG, Salvesen O, Vaag J, Torgersen T. Feasibility, acceptability and preliminary evaluation of a user co-facilitated psychoeducational programme: a feasibility proof-of-concept randomised control trial. BMC Psychiatry. 2024 Sep 16;24(1):615. doi: 10.1186/s12888-024-06015-4. PMID 39285365